CLINICAL TRIAL: NCT01839773
Title: A Randomized, Open-label, Multicenter, Phase 3 Study for Efficacy and Safety Assessment of DHP107 (Oral Paclitaxel) vs. Taxol® in Patients With Metastatic or Recurrent Gastric Cancer After Failure of First-line Chemotherapy With Fluoropyrimidine +/- Platinum
Brief Title: Phase 3 Study to Compare Efficacy and Safety of DHP107 vs. Taxol® in Patients With Metastatic or Recurrent Gastric Cancer
Acronym: DREAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107CS-3
Record Dates: First submitted 2013-04-12; First posted 2013-04-25 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stage IV Gastric Cancer
Keywords: Stomach Neoplasms; Cancer of Stomach; Gastric Cancer; Gastric Neoplasms; Neoplasms, Gastric; Neoplasms, Stomach; Stomach Cancer; paclitaxel; Taxol
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHP107 (oral paclitaxel) (Experimental): DHP107 (oral paclitaxel) will be administered weekly as second line chemotherapy in patients with metastatic or recurrent gastric cancer after failure of first line chemotherapy with fluoropyrimidine +/- platinum.
  Interventions: Drug: Paclitaxel
- Taxol® (IV paclitaxel) (Active Comparator): Taxol® (IV paclitaxel) will be administered 3-weekly as second line chemotherapy in patients with metastatic or recurrent gastric cancer after failure of first line chemotherapy with fluoropyrimidine +/- platinum.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Oral administration on day 1,8,15 of 4-week cycle until progression, unacceptable toxicity or withdrawal of informed concent
  Other Names: DHP107
  Arms: DHP107 (oral paclitaxel)
Drug: Paclitaxel — Premedication, IV infusion on day 1 of 3-week cycle until progression, unacceptable toxicity or withdrawal of informed concent
  Other Names: Taxol®
  Arms: Taxol® (IV paclitaxel)

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of DHP107 (Oral paclitaxel) in comparison to Taxol®(IV paclitaxel) in Patients With Metastatic or Recurrent Gastric Cancer After Failure of 1st Line Chemotherapy With Fluoropyrimidine +/- Platinum.

ELIGIBILITY:
Inclusion Criteria:

1. ≥20 years of age
2. Histologically or cytologically confirmed unresectable, recurrent or metastatic gastric cancer
3. Failure of a first line therapy with fluoropyrimidine +/- platinum for metastatic or recurrent disease.(Adjuvant chemotherapy is not considered as a first line chemotherapy unless recurrence developed within 6 months of completion of adjuvant therapy.)
4. Adequate bone marrow, liver and renal functions
5. INR ≤ 2.0
6. ECOG performance status ≤ 2
7. Neuropathy grade ≤ 1
8. Life expectancy of at least 3 months
9. Measurable lesion according to RECIST version 1.1 on CT scan
10. Written informed consent
11. Patients of child bearing age have to agree to the usage of adequate contraception from before the registration to the study, during the participation period and 90 days after the end of treatment. Female of child bearing age has to show negative for urin pregnancy test within 7 days from beginning of the start of administration. Amenorrhea status has to be sustained for at least 12 months to be considered non-pregnant in case of postmenstrual women.

Exclusion Criteria:

1. Major infectious disease, neurological disorder, or bowel obstruction.
2. Patients with CNS metastases(confirmed through brain imaging if there are symptoms)
3. Patient diagnosed with another cancer type (except non-melanoma skin cancer, cervical cancer, or any other cancer that did not recur or metastasized for more than 5 years and considered as complete remission can be registered)
4. Patient who received radiation therapy within past 2 weeks or who had major surgery including organ resection within past 4 weeks from random assignment date
5. Patient with the history of failure to the taxane chemotherapy
6. Patient who need chronic concomitant use of P glycoprotein, immune suppressor, proton pump inhibitor, or H2-receptor antagonist during the period of clinical trial
7. Chronic treatment using steroid (except oral, local injection, or for externally applied) or other immune suppressor
8. Patient with myocardial infarction, congestive heart failure, arrhythmia showing abrupt change in the ECG, severe or unstable angina, or other serious heart disease
9. Patient with other serious internal disease (chronic obstructive or chronic inhibitory lung disease including shortness of breathe at rest due to all reasons, uncontrollable diabetes and hypertension)
10. History of abuse of a drug or alcohol within 3 months
11. Lactating or pregnant women, or patient (or spouse) who has no intension of using, or cannot use very effective mean of contraception
12. Patient who has or is suspected to have problem in bile acid secretion
13. Patient with active gastrointestinal bleeding, or taking oral anti- vitamine K (With the exception of low dose of Warfarin and acetylsalicylic acide when INR≤2.0)
14. History of serious hypersensitive reaction to the main ingredient or the excipient of the investigational drug
15. History of being seropositive for HIV (HIV test is not a prerequisite).
16. Patients with gastrointestinal dysfunction or on enteral feeding
17. Other patients who are deemed inadequate to participate in the clinical trial by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Participants will be followed until progression, an expected average of 4 months.
  PFS is defined as the time From date of randomization until the date of first documented progression or death, assessed up to 24 months.

SECONDARY OUTCOMES:
Overall Survival | Until 6 months after the last participant is enrolled, assessed up to 24 months.
  OS is defined as the time from the date of inclusion to the date of death, regardless of the cause of death.
Overall Response Rate | Participants will be followed every 6 weeks until progression, an expected average of 4 months.
  ORR is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1) criteria.

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Jungnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Kang YK, Ryu MH, Park SH, Kim JG, Kim JW, Cho SH, Park YI, Park SR, Rha SY, Kang MJ, Cho JY, Kang SY, Roh SY, Ryoo BY, Nam BH, Jo YW, Yoon KE, Oh SC. Efficacy and safety findings from DREAM: a phase III study of DHP107 (oral paclitaxel) versus i.v. paclitaxel in patients with advanced gastric cancer after failure of first-line chemotherapy. Ann Oncol. 2018 May 1;29(5):1220-1226. doi: 10.1093/annonc/mdy055. PMID 29438463